CLINICAL TRIAL: NCT05282823
Title: POLARx™ Cardiac Cryoablation System Post Market Clinical Study POLAR SMART
Brief Title: POLARx™ Cardiac Cryoablation System Post Market Clinical Study (POLAR SMART)
Acronym: POLAR SMART
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PY007
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Subjects: Subjects will be clinically indicated for pulmonary vein isolation ablation procedure (in compliance with instructions for use (IFU)/Tenpubunsyo as legally approved conditions) for the treatment of paroxysmal AF.
  Interventions: Device: Boston Scientific Cardiac Cryoablation System

INTERVENTIONS:
Device: Boston Scientific Cardiac Cryoablation System — is indicated for cryoablation and electrical mapping of the pulmonary veins for pulmonary vein isolation (PVI) in the ablation treatment of AF as per current and future guidelines and system IFU/ Tenpubunsyo.

SUMMARY:
This is a post-market study collecting real-world clinical data on safety, effectiveness and procedural success of Boston Scientific Cardiac Cryoablation System (POLARx™ System)

DETAILED DESCRIPTION:
The study will collect real-world clinical data on safety, effectiveness and procedural success of Boston Scientific Cardiac Cryoablation System (POLARx™ System) when used to perform pulmonary vein isolation (PVI) in the ablation treatment of De Novo Atrial Fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects indicated for the treatment of AF with the cryoablation system;
2. Subjects who are willing and capable of providing informed consent;
3. Subjects who are willing and capable of participating in all testing associated with this clinical study at an approved clinical investigational center;
4. Subjects who are of legal age to give informed consent specific to the national law.

Exclusion Criteria:

1. Any known contraindication to an AF ablation or anticoagulation, including those listed in the IFU/Tenpubunsyo as legally approved conditions;
2. Any prior LA ablation;
3. AF secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause;
4. Known or pre-existing severe Pulmonary Vein Stenosis;
5. Evidence of cardiac myxoma, LA thrombus or intracardiac mural thrombus;
6. Previous cardiac surgery (e.g. ventriculotomy or atriotomy, CABG, PTCA, PCI, ventricular fistula or atrial incision) and any surgery within 90 days prior to enrollment;
7. Any implanted cardiac device (e.g. PM, ICD, CRT, valve replacement, LAAO, etc) within 90 days prior to enrollment;
8. Any planned OR scheduled cardiac device procedure (e.g. PM, ICD, CRT, valve replacement, LAAO, etc) during and post PVI ablation (during and post-index procedure);
9. Any planned ablation in LA except PVI procedure and roof line ablation;
10. Any planned ablation in ventricles;
11. Subjects undergoing atrial septal defect patch or other surgical procedures at or near the atrial septal defect;
12. Subjects with severe valvular disease OR with a prosthetic - mechanical or biological - heart valve (not including valve repair and annular rings);
13. Presence of any pulmonary vein stents;
14. Subjects with active systemic infection;
15. Subjects that have vena cava embolic protection filter devices and/or known femoral thrombus;
16. Any previous history of cryoglobulinemia;
17. Subjects that are unable to undergo atrium access safely or operate in the atrium as per investigator's medical judgement;
18. Subjects with no vascular access or obstruction of the femoral vein;
19. Subjects with blood coagulation disorders or diseases;
20. Any prior history of documented cerebral infarct, TIA or systemic embolism (excluding a post-operative deep vein thrombosis (DVT)) ≤ 180 days prior to enrollment;
21. Subjects who are hemodynamically unstable;
22. The subject is unable or not willing to complete follow-up visits and examination for the duration of the study;
23. Subjects with life expectancy ≤ 1 year per investigator's medical judgement;
24. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (assessment per investigator's discretion);
25. Subjects with unrecovered/unresolved Adverse Events from any previous invasive procedure;
26. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with POLAR SMART study. Exception when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be brought to the attention of the sponsor for approval.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be clinically indicated for PVI ablation procedure (in compliance with instructions for use (IFU)/Tenpubunsyo as legally approved conditions) for the treatment of paroxysmal AF.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Nitta, Principal Investigator — Sakakibara Heart Institute
Locations (19):
- Japan (17):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Chiba University Hospital, Chiba, Chiba
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka-shi, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - National Cerebral and Cardiovascular Center Hospital, Suita-shi, Osaka
  - Saitama Red Cross Hospital, Saitama, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - Sakakibara Heart Institute, Fuchu-shi, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa-shi, Tokyo
  - Kobe City Medical Center General Hospital, Kobe
  - Kobe University Hospital, Kobe
- South Korea (2):
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Subjects
Started | 295
Completed | 276
Not Completed | 19
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 1
Not completed — did not meet protocol criteria | 2
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Includes all treatment subjects
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 193
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 40
  Japan | 253

OUTCOME MEASURES:

1. Primary Outcome: Safety Event Free Rate
Description: Freedom from procedure and device-related adverse events post-index procedure
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 293
Participants | 285

2. Primary Outcome: Failure Free Rate
Description: Failure to achieve acute procedural success during the procedure, or any documented recurrent AF episode(s), or new onset of atrial flutter (AFL) or any other atrial tachycardia (AT) events between Days 91 and 12-Month, or any interventions for AF/AFL/AT between Days 91 and 12-Month
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 293
Participants | 222

3. Secondary Outcome: Failure Free Rate
Description: Failure to achieve acute procedural success during the procedure, or any documented recurrent AF episode(s), or new onset of atrial flutter (AFL) or any other atrial tachycardia (AT) events between Days 91 and 6-Month, or any interventions for AF/AFL/AT between Days 91 and 6-Month
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Subjects
Number analyzed (Participants) | 293
Participants | 236

ADVERSE EVENTS:
Time Frame: Any reportable event, experienced by the study subject after informed consent to 12-month follow-up visit.
Arm/Group | Treatment Subjects
All-Cause Mortality (participants affected / at risk) | 0/293
Serious Adverse Events (participants affected / at risk) | 25/293
Other Adverse Events (participants affected / at risk) | 30/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Subjects (N=293)
AV Block (Transient) (Cardiac disorders) | 1 (1)
Atrial Fibrillation (AF) (Cardiac disorders) | 5 (5)
Atrial Flutter (Cardiac disorders) | 1 (2)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Multiple Heart Failure Symptoms (Cardiac disorders) | 1 (1)
Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 2 (2)
Endocrine (Endocrine disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 3 (3)
Adverse Reaction - Allergic Reaction (General disorders) | 1 (1)
Chest Pain - Other (General disorders) | 1 (1)
Syncope (General disorders) | 1 (2)
Fistula (arterial/venous) (Injury, poisoning and procedural complications) | 1 (1)
Gastroparesis (Injury, poisoning and procedural complications) | 2 (2)
Myocardial Perforation with Tamponade (Injury, poisoning and procedural complications) | 1 (1)
Procedure related Genitourinary/Renal (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Neurological (Nervous system disorders) | 3 (3)
Genitourinary (Renal and urinary disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Subjects (N=293)
EP/Ablation Procedure - Other (Injury, poisoning and procedural complications) | 5 (5)
Esophagitis (Injury, poisoning and procedural complications) | 1 (1)
Fistula (arterial/venous) (Injury, poisoning and procedural complications) | 1 (1)
Gastroparesis (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Pain cardiovascular (non-ischemic) (Injury, poisoning and procedural complications) | 1 (1)
Palpitations (Injury, poisoning and procedural complications) | 1 (1)
Phrenic Nerve Injury Permanent (Injury, poisoning and procedural complications) | 2 (2)
Phrenic Nerve Injury Temporary (Injury, poisoning and procedural complications) | 11 (11)
Procedure related Gastrointestinal (Injury, poisoning and procedural complications) | 2 (2)
Procedure related Genitourinary/Renal (Injury, poisoning and procedural complications) | 2 (2)
Procedure related Pulmonary (including cough, hemoptysis) (Injury, poisoning and procedural complications) | 1 (1)
Neurological (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT05282823/Prot_SAP_000.pdf